CLINICAL TRIAL: NCT01409070
Title: Head to Head Comparison of Azacitidine and Decitabine in Myelodysplastic Syndrome: Retrospective, Multicenter Study
Brief Title: Head to Head Comparison of Azacitidine and Decitabine in Myelodysplastic Syndrome
Acronym: H-1012-015-342
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Inho Kim, Professor, Seoul National University Hospital
Other Study IDs: H-1012-015-342
Record Dates: First submitted 2011-07-28; First posted 2011-08-03 (Estimated); Last update posted 2012-10-16 (Estimated); Status verified 2012-10

CONDITIONS: Myelodysplastic Syndromes
Keywords: MDS
MeSH Terms: conditions — Myelodysplastic Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- Azacitidine: 200 MDS patients taking Azacitidine will be assessed
- Decitabine: 100 MDS patients taking Decitabine will be assessed

SUMMARY:
In Myelodysplastic syndrome, epigenetic treatments such as Azacitidine and Decitabine have been highlighted in phase 3 studies. However, as the 1st line treatment, it has not been evaluated the head to head comparison of two drugs. This study is a retrospective study to compare the efficacy of two drugs.

DETAILED DESCRIPTION:
Among 300 MDS patient, 200 of them have been taking Azacitidine and 100 of them have been taking Decitabine. Medical chart of these patients will be reviewed to assess the efficacy and safety between two agents.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed MDS by bone marrow examination
* Receiving azacitidine and decitabine as a first line chemotherapy
* Adequate hepatic, cardiac, and renal function

Exclusion Criteria:

* Previously treated with another anti-cancer therapy due to MDS
* Not available for clinical information

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: MDS patients who are diagnosed at SNUH
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2011-01; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Response rate | 6 months
  Compare Azacitidine and Decitabine's treatment response rate in MDS patients

SECONDARY OUTCOMES:
Efficacy | 6 months
  To compare hematologic improvement between Azacitidine and decitabine
Survival rate | 6 months
  To compare survival rate between Azacitidine and decitabine
Number of participants with non-hematologic toxicities | 6 months
  To compare toxicity between Azacitidine and decitabine
infection rate | 6 months
  To compare infection rate between Azacitidine and decitabine

CONTACTS AND LOCATIONS:
Locations (1):
- SNUH, Seoul, South Korea

REFERENCES:
- [Derived] Lee YG, Kim I, Yoon SS, Park S, Cheong JW, Min YH, Lee JO, Bang SM, Yi HG, Kim CS, Park Y, Kim BS, Mun YC, Seong CM, Park J, Lee JH, Kim SY, Lee HG, Kim YK, Kim HJ; Korean Society of Haematology AML/MDS working party. Comparative analysis between azacitidine and decitabine for the treatment of myelodysplastic syndromes. Br J Haematol. 2013 May;161(3):339-47. doi: 10.1111/bjh.12256. Epub 2013 Feb 21. PMID 23432512